CLINICAL TRIAL: NCT00969865
Title: Individualized Comprehensive Atherosclerosis Risk-reduction Evaluation Program
Acronym: iCARE
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: iCARE
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individualized Managment Group: Participants receiving, in addition to standard of care, blood tests for markers of heart disease, DNA and RNA analysis, and coronary artery calcium scan.
- Standard Management Group: Participants who receive standard of care.

SUMMARY:
This study will evaluate the effectiveness of an individualized approach to diagnosing and/or treating atherosclerosis. This will be done by combining genetic information, lifestyle information, participant education, and imaging tests to track diagnoses, therapies, and treatment on two groups: 1) Standard Management Group (diagnosed and/or treated according to standard of care) and 2) Individualized Management Group (standard of care plus genetic testing and coronary artery calcium scans).

DETAILED DESCRIPTION:
The purpose of this proposal is to create a large, community-based demonstration project to evaluate the value of a highly individualized approach to atherosclerosis risk reduction. In this project we set out to compare the delivery of appropriate therapies and resource utilization using current national guidelines for the management of atherosclerosis and will compare this to using a highly individualized approach for atherosclerosis risk reduction, based on the evaluation of specific features in individuals and tailoring management based on this evaluation. We plan to show that utilizing the iCARE Program, more patients will receive appropriate diagnoses and subsequent therapies in a more efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* No known coronary artery disease

  * no prior coronary disease by cardiac catheterization (≤39% in any major epicardial vessel)
  * no prior myocardial infarction
  * no prior ST-elevation myocardial infarction (1 mm ST-elevation in 2 contiguous leads)
  * no prior non-ST-elevation myocardial infarction (CK-MB > 2x ULN or elevated troponin that is indicative of myocardial necrosis based on local institutional cutpoints)
  * no prior coronary revascularization procedure
* Intermediate or high Framingham Risk Score (10-year risk 10% or greater)
* Ability and willingness to provide consent and Authorization for use of PHI

Exclusion Criteria:

* Presence of known cardiomyopathy
* Presence of permanent pacemaker, defibrillator, or CRT device
* Presence of clinically significant, uncontrolled arrhythmia (chronic or paroxysmal atrial fibrillation is NOT an exclusion. Arrhythmias treated successfully with ablation are not an exclusion.
* Presence of a known genetic abnormality of cholesterol metabolism (e.g. familial hypercholesterolemia)
* Inability or unwillingness to adhere to follow up schedule
* Inability or unwillingness to provide informed consent and Authorization for use of PHI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with no known coronary artery disease and who have an intermediate or high Framingham Risk Score (10 year risk 10 percent or greater).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of subjects and patients who are diagnosed with subclinical and clinically significant coronary atherosclerosis with the PHI-ACE-iCARE approach, compared to the current guideline-driven approach. | 6 months, 12 months, 18 months

SECONDARY OUTCOMES:
To determine the proportion of patients who receive appropriate revascularization procedures for clinically significant coronary atherosclerosis with the PHI-ACE-iCARE approach, compared to the current guideline-driven approach. | 6 month, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Miller, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States